



#### LEMBAR PENJELASAN KEPADA CALON SUBJEK

Saya, dr. Taufik Mesiano, Sp.S(K) dari bagian Ilmu Saraf Fakultas Kedokteran Universitas Indonesia akan melakukan penelitian dengan judul

"PENGARUH ASUPAN ANTOSIANIN UBI JALAR UNGU TERHADAP VASOMOTOR REACTIVITY PEMBULUH DARAH INTRAKRANIAL PASIEN CEREBRAL SMALL VESSEL DISEASE KAJIAN TERHADAP BHI, L-ARGININE, ADIPONEKTIN, NITRIC OXIDE, FUNGSI KOGNITIF, DAN GAIT".

Saya akan memberikan informasi kepada Bapak/Ibu/Saudara mengenai penelitian ini dan mengundang Bapak/Ibu/Saudara untuk menjadi bagian dari penelitian ini.

Cerebral Small Vessel Disease (CSVD) adalah penyakit pada pembuluh darah kecil di otak akibat adanya sumbatan pada aliran darah. Penyakit ini dapat menyebabkan menurunnya fungsi aktivitas sehari hari, seperti fungsi berfikir dan kemampuan fungsional pada usia lanjut. Berdasarkan penelitian sebelumnya, angka kejadian CSVD dinyatakan tinggi pada penduduk Asia, termasuk Indonesia. CSVD juga terjadi pada usia produktif sebanyak 49,2% (Salim et al., 2018).

Pada penelitian ini Bapak/Ibu/Saudara akan mengonsumsi ekstrak air ubi jalar ungu selama 14 hari. Beberapa pemeriksaan akan dilakukan sebelum (*pre-test*) dan sesudah (*post-test*) konsumsi ekstrak air ubi jalar ungu. Pemeriksaan tersebut adalah USG di bagian kepala, pengambilan darah, pemeriksaan fungsi fikir serta pemeriksaan fungsi berjalan. Prosedur pemeriksaan akan dijelaskan lebih detail oleh Peneliti di setiap sesi. Pada penelitian ini Bapak/Ibu/Saudara juga akan dilakukan pemantauan makanan yang dikonsumsi dalam 24 jam terakhir selama 3 hari oleh peneliti, yaitu pada dua hari kerja (*weekday*) dan satu hari libur (*weekend*).

Antosianin adalah salah satu senyawa yang sering didapatkan dari berbagai tanaman. Ubi jalar ungu merupakan salah satu tanaman yang mengandung antosianin tinggi. Antosianin berperan memberikan warna ungu cerah pada umbi, serta bermanfaat sebagai antioksidan, antidang dan berpotensi fitoestregonik (kandungan dalam tanaman yang fungsinya mirip hormon estrogen di dalam tubuh manusia). Pada beberapa penelitian sebelumnya, antosianin dapat menurunkan resiko obesitas, diabetes, kolesterol tinggi dan menunjukkan potensi dalam meningkatkan fungsi pembuluh darah.

L-Arginin adalah salah satu protein di dalam tubuh yang berfungsi meningkatkan kadar *Nitic Oxide* dan melebarkan pembuluh darah. *Nitric Oxide* adalah senyawa utama yang berperan untuk mempertahankan





FKUI Rumah Sakit Umum Pusa

sirkulasi darah di dalam otak. Adiponektin adalah salah satu senyawa protein yang dihasilkan oleh kelenjar lemak di dalam tubuh yang dapat membantu metabolisme energi pada tubuh. Pada pemeriksaan darah tersebut diharapkan terjadinya peningkatan kadar dalam darah yang menggambarkan ada pelebaran pembuluh darah sehingga membantu penyembuhan pada pasien CSVD. *Trail Making Test* A dan B merupakan salah satu pemeriksaan fungsi fikir dengan menilai kecepatan menyelesaikan soal yang telah diberikan contoh sebelum sesi pengerjaan. Bapak/Ibu/Saudara juga akan melakukan pemeriksaan *Timed Up and Go Test* untuk mengetahui fungsi dan gaya berjalan dengan mengukur waktu berjalan sejauh 3 meter di ruang pemeriksaan, dan berputar balik ke tempat semula sebanyak 3x.

Bapak/Ibu/Saudara dapat berpartisipasi dalam penelitian ini dengan cara menandatangani formulir ini. Jika Bapak/Ibu/Saudara setuju untuk berpartisipasi dalam penelitian ini, Bapak/Ibu/Saudara kapan saja dapat secara bebas mundur dari penelitian ini. Bapak/Ibu/Saudara juga berhak untuk menerima informasi terbaru dari kami mengenai penelitian yang sedang diujikan, jika ada. Jika Bapak/Ibu/Saudara menolak untuk berpartisipasi atau mundur dari penelitian ini, keputusan tersebut tidak akan mempengaruhi hubungan Bapak/Ibu/Saudara dengan saya dan tidak akan berdampak pada pelayanan yang berlaku di rumah sakit ini.

Jika Bapak/Ibu/Saudara tidak memahami setiap pernyataan dalam formulir ini, Bapak/Ibu/Saudara dapat mengajukannya kepada saya.

#### 1. Tujuan penelitian

Tujuan penelitian ini adalah untuk mengetahui efek pemberian ekstrak air ubi jalar ungu terhadap kesehatan pembuluh darah pada pasien CSVD (*Cerebral Small Vessel Disease*).

## 2. Partisipasi dalam penelitian

Dalam kerangka penelitian ini, kami mohon kesediaan Bapak/Ibu/Saudara untuk mengikuti jadwal yang telah kami tetapkan dan memastikan bahwa Bapak/Ibu/Saudara dapat mematuhi jadwal tersebut. Penelitian ini akan melibatkan Bapak/Ibu/Saudara dalam serangkaian kegiatan, termasuk sesi wawancara, pemeriksaan fisik, pemeriksaan saraf, pemeriksaan USG di bagian kepala untuk mengevaluasi pembuluh darah otak, pemberian ekstrak air ubi jalar ungu selama 14 hari, pengisian formulir dan pengisian diari makanan sehari-hari selama penelitian. Kami memperkirakan bahwa waktu yang dibutuhkan akan berlangsung selama 16 hari. Obat yang rutin dikonsumsi tetap dilanjutkan salama penelitian. Peneliti akan mencatat jenis obat yang dikonsumsi beserta dosisnya pada saat wawancara. Penelitian ini akan melibatkan Bapak/Ibu/Saudara dalam beberapa sesi pertemuan oleh dokter. Setiap sesi pertemuan kira-kira akan berlangsung selama 4 sampai 5 jam.





### 3. Alasan memilih Bapak/Ibu/Saudara

Pemilihan peserta pada penelitian ini dilakukan berdasarkan aturan yang sudah ditetapkan. Hal ini dilakukan dengan tujuan untuk memastikan bahwa peserta yang terlibat memiliki karakteristik yang sesuai dengan tujuan penelitian, sehingga tanggapan terhadap ekstrak air ubi jalar ungu dapat lebih akurat dan relevan.

Kriteria masuk untuk penelitian ini termasuk rentang usia antara 40-65 tahun, kemampuan serta kesediaan untuk mengikuti seluruh tahapan penelitian hingga selesai, dan kesediaan untuk menandatangani lembar persetujuan informasi (*informed consent*). Selain itu, peserta dalam kelompok ini juga diharapkan memiliki kemampuan kognitif yang memadai, serta memiliki kemampuan berjalan mandiri.

#### 4. Prosedur Penelitian

- Setelah menyetujui dan menandatangani formulir ini, Anda akan diwawancarai oleh dokter untuk menanyakan: Identitas diri, riwayat penyakit, riwayat penggunaan obat, riwayat alergi, riwayat konsumsi suplemen herbal atau multivitamin, kebiasaan minum minuman keras atau minum minuman yang mengandung alkohol.
- Anda akan menjalani pemeriksaan fisik umum, pemeriksaan neurologis, serta pemeriksaan USG kepala oleh peneliti untuk keperluan skrining penelitian.
- 3. Jika Anda telah memenuhi kriteria yang telah ditetapkan oleh peneliti, maka akan diikutsertakan ke tahap penelitian selanjutnya.
- 4. Semalam sebelum hari pertama penelitian (mulai pukul 21.00), Anda diminta berpuasa, namun diperbolehkan minum air putih seperlunya.
- 5. Pada hari pertama dimulainya penelitian, Anda diminta datang pada pukul 07.00 untuk selanjutnya dilakukan pengambilan darah.
- 6. Pengambilan darah dilakukan dengan cara memasang jarum kupu-kupu pada pembuluh darah di lengan bawah. Pengambilan darah dilakukan melalui jarum kupu kupu yang sudah dipasang. Pengambilan darah sebanyak kira-kira dua sendok makan dan satu sendok teh. Efek samping yang mungkin akan terjadi yaitu nyeri di bekas suntikan atau perdarahan dan memar yang dapat hilang seiring dengan waktu. Efek samping yang lebih serius dapat berupa infeksi dan perdarahan yang berlebih, namun efek tersebut jarang terjadi. Semua efek samping yang terjadi dapat diinformasikan kepada tim peneliti untuk penanganan lebih lanjut.
- 7. Pengambilan darah pertama ini untuk pemeriksaan laboratorium mengenai keadaan darah yaitu darah lengkap, fungsi ginjal, fungsi hati, gula darah sewaktu, serta parameter darah khusus yang telah dijelaskan sebelumnya (*Nitric Oxide, L-arginine, adiponectin, dan antosianin*).
- 8. Pengambilan darah dilakukan oleh perawat yang sudah terbiasa mengambil darah.
- 9. Kemudian dilanjutkan dengan pemeriksaan fungsi fikir, fungsi berjalan dan USG di bagian kepala.





FKUI Rumah S

- 10. Pada pemeriksaan fungsi fikir, Anda akan mengerjakan 2 lembar kertas berupa soal dengan mengurutkan angka dan huruf. Pada setiap lembar, tim peneliti akan memberikan contoh cara penyelesaian soal terlebih dahulu. Waktu penyelesaian soal akan dicatat saat pertama kali tim peneliti mengatakan "Mulai" dan diakhiri sampai pada angka atau huruf terakhir yang dikerjakan.
- 11. Pada pemeriksaan fungsi berjalan, Anda akan berada di dalam ruangan dengan luas 3 x 5meter dan berjalan sebanyak 3x. Awalnya, Anda akan duduk di kursi yang telah disediakan, kemudian berdiri dan berjalan sejauh 3meter sesuai tanda yang telah diberikan dan berputar balik untuk duduk kembali. Peneliti akan memberikan contoh terlebih dahulu. Pada pemeriksaan ini akan dicatat waktunya sejak pertama kali peneliti mengatakan "Go" dan diakhiri sampai Anda duduk di kursi kembali.
- 12. Pemeriksaan USG kepala dilakukan oleh Dokter Spesialis Saraf/Peneliti yang memiliki keahlian khusus dalam bidang neurosonologi. Saat menjalani pemeriksaan, Anda akan berbaring di tempat tidur pemeriksaan, teropong USG ditempatkan di bagian samping kepala, dekat dengan daerah pelipis atau sekitar telinga. Anda akan merasakan tekanan ringan dari alat yang ditempelkan, namun tidak ada rasa nyeri. Nilai reaksi dari pembuluh darah otak yang diteliti akan diperoleh pada saat Anda menahan nafas selama 30 detik kemudian dibandingkan dengan saat bernafas biasa.
- 13. Setelah serangkaian pemeriksaan awal (pre-test) selesai, Anda akan menerima pemberian asupan antosianin dari ekstrak air ubi jalar ungu sebanyak 500mL per hari, dengan pemberian dua kali sehari (masing-masing 250 mL dalam 1 botol) yang akan diberikan oleh peneliti selama 14 hari berturutturut.
- 14. Anda akan dihubungi oleh tim peneliti untuk memantau makanan yang dikonsumsi 24 jam terakhir selama 3 hari, yaitu pada dua hari kerja (*weekday*) dan satu hari libur (*weekend*) pada minggu pertama dan kedua.
- 15. Pada hari ke 16 penelitian, semalam sebelum pemeriksaan (mulai pukul 21.00), Anda diminta berpuasa, namun diperbolehkan minum air putih seperlunya.
- 16. Pada hari evaluasi penelitian, Anda diminta datang pada pukul 07.00 untuk selanjutnya dilakukan pengambilan darah yaitu darah lengkap, fungsi ginjal, fungsi hati, gula darah sewaktu, serta parameter darah khusus yang telah dijelaskan sebelumnya (*Nitric Oxide, L-arginine, adiponectin, dan antosianin*).
- 17. Kemudian dilanjutkan dengan pemeriksaan fungsi fikir, fungsi berjalan dan USG kepala seperti yang telah dilakukan saat pemeriksaan awal (pre-test).

### 5. Risiko, efek samping dan tatalaksananya

Dalam rangka menjaga keselamatan dan kenyamanan peserta, telah diambil langkah-langkah pencegahan yang ketat dengan menerapkan proses pengolahan yang higienis dalam penelitian ini. Walaupun demikian, penting





untuk diingat bahwa terdapat potensi risiko yang perlu diperhatikan, terutama terkait dengan kemungkinan reaksi alergi terhadap ekstrak air ubi jalar ungu, terutama bagi individu yang memiliki sensitivitas tertentu.

Selain risiko tersebut, perlu juga mempertimbangkan kemungkinan adanya efek samping seperti gangguan pencernaan, seperti mual atau gangguan perut ringan akibat konsumsi ekstrak tersebut. Aspek ini akan diawasi dengan cermat selama penelitian guna memastikan keselamatan dan kenyamanan peserta. Apabila Bapak/Ibu/Saudara mengalami efek samping atau gangguan tersebut, tim penelitian telah siap untuk memberikan tatalaksana yang sesuai dan, bila perlu, merujuk Bapak/Ibu/Saudara untuk mendapatkan perawatan medis lebih lanjut.

Tim peneliti akan melakukan pemantauan yang teliti terhadap reaksi dan efek samping selama seluruh periode penelitian. Apabila terjadi reaksi alergi atau efek samping yang serius, Bapak/Ibu/Saudara akan segera dirujuk untuk mendapatkan konsultasi medis lebih lanjut. Jika timbul efek samping atau risiko yang signifikan, partisipasi Bapak/Ibu/Saudara dalam penelitian ini dapat dihentikan demi menjaga kesejahteraan dan keselamatan Bapak/Ibu/Saudara.

#### 6. Manfaat

Partisipasi Bapak/Ibu/Saudara akan memberikan kontribusi positif terhadap pengembangan pangan fungsional yaitu antosianin dari ekstrak air ubi jalar ungu terhadap kesehatan pembuluh darah pasien CSVD. Pemeriksaan fisik, mencakup tanda-tanda vital, kognitif, pemeriksaan berjalan, evaluasi pembuluh darah otak, dan pemeriksaan laboratorium darah akan memberikan informasi penting mengenai kondisi kesehatan Bapak/Ibu/Saudara. Hal ini membantu Bapak/Ibu/Saudara untuk memantau kesehatan pribadi, mendapatkan pemahaman yang lebih mendalam, serta mengidentifikasi potensi masalah kesehatan yang perlu ditangani lebih lanjut.

### 7. Kompensasi

Apabila Bapak/ibu/saudara telah memenuhi kriteria sampel penelitian dan akan menjalankan pre test, maka Bapak/ibu/saudara mendapatkan uang ganti transportasi sebesar [Rp 150.000]. Dan apabila Bapak/ibu/saudara telah melaksanakan penelitian dengan mengonsumsi ekstrak air ubi jalar ungu selama 14 hari, maka akan mendapatkan kembali uang ganti transportasi untuk pemeriksaan post test sebesar [Rp 150.000].

### 8. Pembiayaan

Semua biaya yang terkait dengan penelitian ini akan ditanggung oleh pihak peneliti.





#### 9. Kerahasiaan

Seluruh informasi yang terkait dengan identitas subjek penelitian akan dijaga kerahasiaannya dan hanya akan diakses oleh peneliti dan staf penelitian. Hasil dari penelitian ini akan dipublikasikan tanpa mencantumkan identitas subjek penelitian.

### 10. Kewajiban subyek penelitian

Sebagai subjek penelitian, Bapak/Ibu/Saudara diharapkan untuk mematuhi aturan dan petunjuk penelitian sebagaimana yang telah dijelaskan di atas. Jika terdapat hal-hal yang masih belum jelas atau memerlukan penjelasan lebih lanjut, Bapak/Ibu/Saudara dianjurkan untuk mengajukan pertanyaan kepada peneliti.

#### 11. Hak untuk menolak dan mengundurkan diri

Bapak/Ibu/Saudara memiliki kebebasan untuk memilih apakah akan berpartisipasi atau tidak dalam penelitian ini. Persetujuan untuk berpartisipasi tidak diwajibkan, dan Bapak/Ibu/Saudara berhak untuk menarik diri setiap saat. Keputusan ini tidak akan berdampak pada hubungan Bapak/Ibu/Saudara dengan kami maupun layanan di rumah sakit.

#### 12. Akses pasca penelitian (Post-trial access)

Pada akhir penelitian ini, kami akan tetap memberikan Bapak/Ibu/Saudara pengobatan terbaik lanjutan terhadap penyakit Bapak/Ibu/Saudara saat ini sesuai hasil uji.

#### 13. Informasi Tambahan

Bapak/Ibu/Saudara diberikan kesempatan untuk mengajukan pertanyaan terkait penelitian ini agar semua hal yang belum jelas dapat dipahami dengan baik. Apabila terjadi efek samping atau Bapak/Ibu/Saudara memerlukan penjelasan lebih lanjut kapan saja, silakan menghubungi penanggung jawab penelitian, yaitu: Dr. Taufik Mesiano, Sp.S(K), di nomor 081781134.





## LEMBAR PERSETUJUAN KEIKUTSERTAAN DALAM PENELITIAN

| Sertifikat Persetujuan (Consent) | |
|---|---|
| Saya telah membaca semua penjelasan tentang | Saya mengkonfirmasi bahwa peserta telah |
| penelitian ini. Saya telah diberikan kesempatan | diberikan kesempatan untuk bertanya |
| untuk bertanya dan semua pertanyaan saya telah | mengenai penelitian ini, dan semua |
| dijawab dengan jelas. Saya bersedia untuk<br>berpartisipasi pada studi penelitian ini dengan | pertanyaan telah dijawab dengan benar.<br>Saya mengkonfirmasi bahwa persetujuan |
| sukarela. | telah diberikan dengan sukarela. |
| outai ou | totan arooman aongan sanarota. |
| Nama ankial/mali | Nama namaliti/naminta namatainan |
| Nama subjek/wali | Nama peneliti/peminta persetujuan |
| Tanda tangan peserta studi | Tanda tangan peneliti/peminta persetujuan |
| Tanggal | Tanggal |
| hari/bulan/tahun | hari/bulan/tahun |

Semua penjelasan tersebut telah disampaikan kepada saya dan semua pertanyaan saya telah dijawab oleh **dr. Taufik Mesiano, Sp. S (K)**. Saya mengerti bahwa bila memerlukan penjelasan, saya dapat menanyakan kepada **dr. Taufik Mesiano, Sp. S (K)**. Informasi Peneliti:

Peneliti Utama: dr. Taufik Mesiano, Sp. S (K)

No. telp 0817-811-344; email taufik.mesiano@ui.ac.id

KEPK FKUI-RSCM: Jalan Salemba 6, Jakarta Pusat, 10430

No. Telp: 021 3157008 Email: ec\_fkui@yahoo.com